CLINICAL TRIAL: NCT03044392
Title: Determination of the Optimal "Next Bolus" Interval for Programmed Intermittent Bolus Epidural Analgesia: A Randomized Controlled Trial
Brief Title: Determination of the Optimal "Next Bolus" Interval for Programmed Intermittent Bolus Epidural Analgesia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Allana, Anesthesiologist, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1021552
Record Dates: First submitted 2017-01-23; First posted 2017-02-07 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Labor Pain
Keywords: Programmed Intermittent Epidural Bolus; Labour Analgesia; Pain
MeSH Terms: conditions — Labor Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Next Bolus Interval 15 minutes (Active Comparator): Next Bolus Interval 15 minutes
  Interventions: Other: Next Bolus Interval
- Next Bolus Interval 30 minutes (Active Comparator): Next Bolus Interval 30 minutes
  Interventions: Other: Next Bolus Interval
- Next Bolus Interval 45 minutes (Active Comparator): Next Bolus Interval 45 minutes
  Interventions: Other: Next Bolus Interval

INTERVENTIONS:
Other: Next Bolus Interval — Next Bolus Interval 15, 30, or 45 minutes
  Other Names: Time from start of epidural pump to first dose of medication

SUMMARY:
The current standard of practice for the maintenance of epidural analgesia is through use of a continuous infusion pump. Enhanced technology now supports the use of programmed intermittent bolus (PIEB) administration. This novel drug delivery system provides small boluses of local anesthetic and opioid at programmed intervals. Several studies suggest that administration of PIEB allows a more extensive spread of local anesthetic in the epidural space and provides superior labour analgesia compared to traditional continuous epidural infusions. PIEB is associated with lower anesthetic consumption, a shorter second stage of labour and greater patient satisfaction.

The authors are focusing on a PIEB setting known as the "Next Bolus". "Next Bolus" (NB) determines when the first PIEB bolus is given after the initiation of the epidural and starting the PIEB pump. Currently we set this to be 15-45 minutes. In an attempt to optimize resources, authors hope to determine the optimal NB interval that will provide adequate analgesia but limit overall drug consumption. An optimally timed next bolus should minimize drug costs and limit nurse and physician intervention by decreasing the need for manual boluses.Increased local anesthetic consumption can cause undesirable side effects such as itchiness, decreased blood pressure and motor blockade. By assigning patients to receive the NB at 15, 30 or 45 minutes the authors hope to find the interval that provides analgesia while minimizing side effects, improving patient safety. If the bolus is given too late then there may be increased pain, less patient satisfaction, and the need for more analgesia in the form of Patient Controlled Epidural Anesthesia or a manual bolus.The authors hope that determining the NB will result in an institutional change to improve patient outcomes and facilitate knowledge transfer. This information will be the first available research to help guide other obstetrical centres using PIEB technology in determining the optimal NB interval.

DETAILED DESCRIPTION:
Background

Enhanced epidural pump technology now supports the use of automated or programmed intermittent bolus (PIB) administration. Anesthesiologists can now program pumps to deliver small, regularly timed intermittent boluses for maintenance of labour analgesia and specify "lockout" intervals to ensure patient safety.

Several studies suggest that administration of PIB may result in a more extensive spread of local anesthetic in the epidural space and provide superior labour analgesia compared to CEI. In a recently published systematic review by George et al. (1), PIB was associated with lower anesthetic consumption, a shorter second stage of labour and greater patient satisfaction compared to CEI (1).

The optimal PIB volume and dosing interval for programmed intermittent bolus has not been determined. A small volume with a short bolus interval may be associated with similar drawbacks as continuous infusion, while a large volume bolus interval may be associated with increased breakthrough pain and reduced patient satisfaction. Wong et al. showed that extending the PIB interval from 15 min to 60 min with a larger PIB volume (10 mL vs. 2.5 mL) results in decreased anesthetic consumption without affecting patient satisfaction (3). Until recently, there was not a pump that could provide PIB along with PCEA. Smith Medical now produces the CADD pump with this feature. It ensures that that there are specific limits set to not allow "stacking" of boluses and potentially unsafe administration of local anesthetics. This pump now has more variables to program and determine the quality of labour analgesia.

A variable that has not received any research attention is the "Next Bolus" (Figure 5). "Next Bolus" (NB) determines when the first PIB bolus is given after the initiation of the epidural and starting of the pump. Currently we set this to be 15-45 minutes depending on the clinician. Determining the optimal timing of the NB is important because if the bolus is given too late there may be increased pain and less patient satisfaction. This could lead to earlier initiation of PCEA, more frequent PCEA attempts and possibly the need for physician intervention for a manual bolus. As more local anesthetic is delivered, the patient may have a decrease in blood pressure or greater motor blockade (i.e. leg weakness) than desired.

Design & Procedure Potential participants will be identified by research personnel by communicating with the attending anesthesiologist on the Birth Unit and the Clinical Leader of Operations for the Birth Unit at the IWK Health Centre. Birth Unit nurses will receive an educational session and training provided by the research coordinator prior to study commencement. Birth unit nurses will be notified by the Clinical Leader of Operations if their patient meets study inclusion criteria. The patient's nurse will review options for labour pain relief with the patient. These options include non-pharmacological measures (baths, massage, hypnosis etc.), inhaled nitrous oxide, opioid injections, or an epidural. When labour pain management options are introduced, the nurse will provide the patient with a brochure that includes basic study information. If an epidural is requested for labour analgesia, nurses who have received education regarding the study, will ask the patient if they would be willing to speak with research staff. With their consent, participants will be approached by study personnel and informed, written consent will be obtained. As standard care in the birth unit, upon request of labour analgesia, the cervix will be measured and a baseline pain score and blood pressure will be determined.

A staff anesthesiologist will use a combined spinal-epidural (CSE) technique to initiate labour analgesia. As per standard practice at the IWK, an IV catheter will be in place before initiation of the technique. With the patient in the sitting position, the epidural space will be identified at the L3-4 or L2-3 interspace with a 17G, 9 cm Tuohy epidural needle using a loss of resistance to air or saline (< 1 mL) technique. A 27G, 12 cm Whitacre spinal needle will be placed into the shaft of the epidural needle and the presence of cerebrospinal fluid in the hub of the spinal needle will confirm dural puncture. Bupivicaine 0.25% 0.8 mL (2 mg) + Fentanyl 10 mcg (total 1 mL) will be injected into the intrathecal space.

Each participant will be randomly allocated (using a computer generated randomization table) to one of three groups. Group assignments will be sealed in sequentially numbered envelopes that will be opened by study personnel following the consent process. The pump will be programmed by an unblinded member of the anesthesia team (anesthesiologist or anaesthesia assistant) and maintenance epidural analgesia will be initiated in accordance with IWK policies when the epidural procedure is complete. The individual programming the pump will not be collecting data. The start time of the pump will be recorded on the envelope and the sealed envelope will be given to the study personnel. The pump will be connected and initiated once the epidural procedure is complete and will start the infusion exactly 5 minutes after the intrathecal injection. Each participant will have the same PIB settings (PIB bolus 8 mL, PIB interval 45 minutes). Group A will be assigned a NB of 15 minutes, group B 30 minutes and group C 45 minutes.

The data collection will take place in the patient's assigned labour room in the IWK Birth Unit. The CADD Solis Ambulatory Infusion System (Smiths Medical ASD, Inc., St Paul MN) will be used to administer the programmed intermittent epidural bolus doses and patient-controlled epidural analgesia (PCEA). The current IWK labour analgesia standard ensures each labour room is equipped with a Smith Medical CADD pump, epidural infusion tubing and an epidural procedure tray. No new or additional supplies or personnel will be required for the study. Prior to study commencement, the research assistant will be trained by one of the investigators (anesthesiologist) on how to complete a dermatome sensory evaluation and Bromage score. In addition, the research assistant will receive training from the anesthesiologist regarding how to instruct patients to use the PCEA device. For all groups the PCEA will remain standardized. If after two confirmed PCEA doses that participant's pain is not suitably controlled the anesthesiologist will be consulted to provide a manual bolus (0.1% ropivacaine 10 mL). The patient and research personnel recording data will be blinded to the group assignment.

Data to be collected Demographic data and health history Medical record number, maternal age, height, weight, BMI.

Labour Information Gestational age, cervical dilation at initiation of CSE analgesia, duration of labour (initiation of analgesia to delivery), maximum oxytocin infusion rate during labour, mode of delivery, time from initiation of analgesia to delivery.

Analgesia Data Maintenance epidural solution volume administered from programmed intermittent bolus pump, time of first administered PCEA bolus request, number of PCEA bolus requests and delivered doses, PCEA ropivacaine dose, time to first request for manual bolus, number of manual bolus doses, manual bolus ropivacaine dose, total ropivacaine dose, highest thoracic dermatome sensory level to pin prick at 0, 15, 30, 45, 60, 120, 180, 240, 300, and 360 minutes, along with a modified Bromage score, hypotension, need for vasopressors.

Satisfaction Scores Overall maternal satisfaction scores (NRS) will be sought within one day of delivery. Patients will be asked "On a scale from 0 to 100, how satisfied were you with the pain control provided by the epidural during your labour?"

Data Collection In keeping with CONSORT guidelines all participants enrolled will be included in an intention to treat analysis. Descriptive statistics will be expressed as mean +/- standard deviation. The Student's t-test will be used for comparison of the means of continuous, normally distributed data. Two-way ANOVA or Friedman test will be used for variable differences in groups, and Bonferroni or Tukey HSD test will be used for multiple comparisons. Categorical data are to be analyzed using χ2 test or Fisher's exact test, as appropriate. The investigators will perform the statistical analysis, with the assistance of collaborating statistician. An interim analysis will not be conducted and α set at 0.05 for significance. A sample size of 26 per group will have an 80 % power to detect a reduction in the time to first administered PCEA request by 20 minutes at alpha=0.05. To account for any dropouts, we will aim to recruit 35 patients per group.

ELIGIBILITY:
Inclusion Criteria:

* • American Society of Anesthesiologists (ASA) Physical Status I-II (ASA I - Healthy, ASA II - mild and controlled systemic disease)

  * Spontaneous labour
  * Nulliparous parturient
  * Single gestations ≥ 36 weeks
  * English speaking
  * Age 18-45 years
  * Vertex presentation
  * Requesting an epidural for labour analgesia
  * Cervical dilation less than 2 cm or greater than 6 cm at the time of initiation of neuraxial analgesia

Exclusion Criteria:

* • Use of IV opioids within 1 hour of initiating the epidural

  * Use of nitrous oxide after initiating the epidural pump
  * Contraindications to neuraxial analgesia (i.e. coagulopathy, infection, neuropathy)
  * Abnormal spinal anatomy (i.e. scoliosis, spina bifida, spinal instrumentation)
  * Height < 5'0" or BMI ≥ 40 kg/m2
  * Chronic analgesics
  * Diseases of pregnancy (i.e. hypertension, preeclampsia, gestational diabetes)
  * Severe maternal cardiac disease
  * Known fetal anomalies /intrauterine fetal demise
  * Physical or psychiatric condition which may impair cooperation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant
Enrollment: 84 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Time to first administered Patient Controlled Epidural Analgesia (PCEA) request | 360 minutes
  The time from the start of the epidural pump to the first administered request for a PCEA bolus (in minutes).

SECONDARY OUTCOMES:
Pain scores | 360 minutes
  Pain Scores (NRS 0-10) - measured at baseline, 0, 15, 30, 45, 60, 120, 180, 240, 300, and 360 minutes.
Number of PCEA bolus attempts | 360 minutes
  The number of times the patient presses a button requesting a PCEA bolus in the first 360 minutes or until delivery.
Number of PCEA bolus received | 360 minutes
  The number of PCEA boluses actually administered by the pump in the first 360 minutes or until delivery.
Number of manual bolus doses administered by the anesthesiologist | 360 minutes
  The number of times an anesthesiologist had to administer a manual bolus because pain was inadequately controlled with PCEA in the first 360 minutes or until delivery.
Total local anesthetic consumption after pump initiation | 360 minutes
  mg of ropivicaine 0.1% calculated by the CADD pump in the first 360 minutes or until delivery.
Highest thoracic dermatome sensory level | 360 minutes
  Measured by pin-prick at 15, 30, 45, 60, 120, 180, 240, 300, and 360 minutes.
Modified Bromage scores measured at 60, 120, 180, 240, 300, and 360 minutes | 360 minutes
  Measures motor blockade, recorded at 0, 15, 30, 45, 60, 120, 180, 240, 300, and 360 minutes
Maternal satisfaction with labour analgesia | 360 minutes
  0-100%, measured within 24 hours of delivery.
Occurrence of hypotension | 360 minutes
  Defined as a 20% drop of blood pressure from baseline. Measured at baseline, 0, 15, 30, 45, 60, 120, 180, 240, 300, and 360 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Allana Munro, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No